CLINICAL TRIAL: NCT04460599
Title: Description of neurolOgical Involvement Observed During SARS COV2 Infection
Brief Title: Neurological Features During COVID19
Acronym: NeuroSARS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, david orlikowski, Professor, Centre d'Investigation Clinique et Technologique 805
Other Study IDs: Brain COVID
Record Dates: First submitted 2020-07-06; First posted 2020-07-07 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Encephalitis
Keywords: Cranial nerves; brainstem; dysautonomia
MeSH Terms: conditions — Encephalitis; Autonomic Nervous System Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — Observation of recorded neurological signs

SUMMARY:
Description of the neurological impairment: clinico-radiological and electrophysilogical correlations

DETAILED DESCRIPTION:
Describe short and long term clinical radiological and electrophysilogical presentations of neurological damage central and peripheral SARS COV2 infection Describe the association between neurological, respiratory and dysautonomic Determine the prognosis of neurological damages to short and long term.

ELIGIBILITY:
Inclusion Criteria:

* PCR SARS COV2 positive or CT Scan
* Central neurological signs such as confusion, epilepsy, abnormal movement, pyramidal signs, motor or sensory deficit, involvement of cranial pairs (such as anomie or ageusia) or peripheral.
* Dysautonomic signs such as hypotension or hypertension, bradycardia or tachycardia, hypothermia, SIADH not explained by therapy or a pathology other than SARS COV 2 infection

Exclusion Criteria:

* Contraindication to performing an MRI scan
* Minor
* Pregnant woman
* No follow-up possible at 6 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Population hospitalized in ICU for COVID 19.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-03-08 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary | 6 months
  incidence of objective neurological damage

SECONDARY OUTCOMES:
Secondary | 6 months
  incidence of clinical neurological damage incidence of radiological neurological damage incidence of neurophysiological neurological damage

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Raymond Poincare, Garches, France

IPD SHARING:
Plan to Share IPD: No